CLINICAL TRIAL: NCT05620017
Title: A Multicenter, Open Phase I Clinical Study to Evaluate the Safety, Tolerance, Pharmacokinetics and Initial Efficacy of BAT8008 for Injection in Patients With Advanced Solid Tumor
Brief Title: Evaluate the Safety, Tolerability and Pharmacokinetic Characteristics of BAT8008 for Injection
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BAT-8008-001-CR
Record Dates: First submitted 2022-10-25; First posted 2022-11-17 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- A/0.8mg/kg (Experimental): Drug：BAT8008 for Injection,0.8mg/kg
  Interventions: Drug: BAT8008 for Injection
- B/1.2mg/kg (Experimental): Drug：BAT8008 for Injection,1.2mg/kg
  Interventions: Drug: BAT8008 for Injection
- C/2.4mg/kg (Experimental): Drug：BAT8008 for Injection,2.4mg/kg
  Interventions: Drug: BAT8008 for Injection
- D/3.6mg/kg (Experimental): Drug：BAT8008 for Injection,3.6mg/kg
  Interventions: Drug: BAT8008 for Injection
- E/4.8mg/kg (Experimental): Drug：BAT8008 for Injection,4.8mg/kg
  Interventions: Drug: BAT8008 for Injection
- F/6.0mg/kg (Experimental): Drug：BAT8008 for Injection,6.0mg/kg
  Interventions: Drug: BAT8008 for Injection
- G/7.2mg/kg (Experimental): Drug：BAT8008 for Injection,7.2mg/kg
  Interventions: Drug: BAT8008 for Injection

INTERVENTIONS:
Drug: BAT8008 for Injection — Intravenous infusion, once every 2 weeks (Q2W). It is recommended that the infusion time of the first cycle should be ≥ 3 hours. If no infusion reaction occurs, the subsequent circulation can be completed within 1-2 hours.
  Other Names: Recombinant humanized anti Trop2 monoclonal antibody for injection Exetecan conjugate

SUMMARY:
Objectives:To evaluate the safety and tolerability of BAT8008 for injection in patients with advanced solid tumors, explore the maximum tolerated dose (MTD), and provide the recommended dose for subsequent clinical trials.

DETAILED DESCRIPTION:
In this multi-center, open, dose-increasing, dose-expanding Phase I clinical study, rapid titration and a "3+3" dose-increasing design were used to explore the safety, tolerability and PK characteristics of BAT8008 for injection in patients with advanced solid tumors. During the dose-escalation test, appropriate doses were selected for the extended study according to the previous study data.

ELIGIBILITY:
Inclusion Criteria:

All of the following items could be meet to be enrolled the study

1. Age ≥18 years old, both sexes;
2. Voluntarily sign the informed consent;
3. Patients with advanced or metastatic epithelial-derived solid tumors that have been histopathologically or cytologically confirmed, have failed or not been treated with standard therapy, have been intolerant to or have refused standard therapy.
4. According to RECIST1.1, there is at least one measurable tumor lesion;
5. The Eastern Collaborative Oncology Group (ECOG) Performance Status score requires a score of 0 or 1;
6. Investigators assessed the expected survival of ≥12 weeks;
7. Adequate organ and bone marrow reserve function
8. Fertile female patients willing to use effective birth control/contraception to prevent pregnancy during the study period. Male patients must consent to use an effective method of contraception during the study;
9. Willing to provide previously archived or fresh tumor tissue samples
10. Able to understand the test requirements, willing and able to comply with the test and follow-up procedures.

Exclusion Criteria:

If you meet any of the following items, you will not be allowed to enroll this study :

1. Within 4 weeks before the first administration of the study drug, he has received experimental drug treatment or participated in clinical research of medical devices;
2. Have received other anti-tumor treatment within 4 weeks before the first administration of the study drug, such as chemotherapy, radiotherapy (palliative radiotherapy should be completed within 2 weeks before the first administration), targeted therapy/immunotherapy (at least 4 weeks or at least 5 half-life, whichever is shorter), hormone therapy (except alternative therapy);
3. Within 2 weeks before the first administration of the study drug, he has received the treatment of traditional Chinese medicine, Chinese patent medicine or immunomodulatory drugs (including thymosin, interferon, interleukin, etc.) with anti-tumor effect;
4. Before the first administration of the study drug, AE (CTCAE5.0) caused by previous anti-tumor treatment was still greater than grade 1, except for the following conditions: a. alopecia; B pigmentation; c. The distal toxicity caused by chemotherapy and radiotherapy can not be further recovered after judgment;
5. Major surgery (excluding the operation for diagnosis) is required within 4 weeks before the first administration of the study drug or is expected to be performed during the study period;
6. Patients who have received Trop2 targeted therapy previously;
7. Those who have received the treatment containing exatecan or irinotecan and other topoisomerase I inhibitor drugs in the past and have experienced drug related AE ≥ grade 3 or treatment failure of topoisomerase I inhibitor;
8. Have a history of allograft cell or solid organ transplantation;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | At the end of Cycle 1( first cycle is 21 days, subsequent cycles are 14 days)
  DLT was defined as grade 3 or higher toxicity associated with the investigational product that occurred within 21 days of the subject's initial administration
Maximum tolerated dose (MTD) | At the end of Cycle 1( first cycle is 21 days, subsequent cycles are 14 days)
  MTD was defined as exploration in a dose group observed ≤1/6 of subjects during the DLT evaluation period to the highest dose level of DLT.

SECONDARY OUTCOMES:
AUC(0-inf)after cycle 6 administration | 91 days after first dose of BAT8008
  The area under the concentration-time curve extrapolated from time 0 to infinity

OTHER OUTCOMES:
Presence of ADA/nentralizing antibodies（NAbs） | 91 days after first dose of BAT8008
  presence of anti-drug antibody/ nentralizing antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Weier Song, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (2):
- China (2):
  - Affiliated Cancer Hospital of Chongqing University, Chongqing, Chongqing Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang